CLINICAL TRIAL: NCT06201650
Title: Performance of Serum Neurofilament Light Chain in a Wide Spectrum of Clinical Courses of Amyotrophic Lateral Sclerosis - a Cross-sectional and Longitudinal Multicenter Study
Brief Title: Neurofilament Light Chain in Amyotrophic Lateral Sclerosis
Acronym: NfL-ALS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Boris Canessa ALS Stiftung (Unknown)
Responsible Party: Principal Investigator, Thomas Meyer, MD, Prof. Dr. Thomas Meyer, Charite University, Berlin, Germany
Other Study IDs: NfL-ALS
Record Dates: First submitted 2023-04-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: ALS; Amyotrophic lateral sclerosis; Neurofilament light chain; NfL; ALS Funktional Rating Scale; Progression; biomarker; treatment marker; therapeutic marker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Charcot-Marie-Tooth disease, Type 1F; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neurofilament light chain — Neurofilament light chain as biomarker for amyotrophic lateral sclerosis

SUMMARY:
This study assesses the performance of serum neurofilament light chain (sNfL) in amyotrophic lateral sclerosis (ALS) in a wide range of disease courses, in terms of ALS progression, disease duration, and tracheostomy invasive ventilation (TIV). The aim of the research project is to investigate the correlation between NfL serum concentration and the natural course of the disease, the ALS progression rate, and specific phenotypes of ALS. Furthermore, the performance of NfL as a therapeutic biomarker will be studied. A systematic analysis of the NfL serum concentration in a cohort of 3,000 ALS patients using the Single Molecule Analysis method (SIMOA) will be performed. This analysis is carried out as a multi-center study.

DETAILED DESCRIPTION:
The aim of this study is to investigate the correlation between the NfL serum concentration and the natural course of the disease, the ALS progression rate as measured by the ALS functional rating scale (ALSFRS-R), and specific phenotypes of ALS. The results of the study will contribute to the assessment of disease progression and the prognosis making of ALS. Furthermore, the performance of NfL as a therapeutic marker of ALS medicines and non-pharmacologic treatment options will be investigated. A systematic analysis of the NfL serum concentration in an extended cohort of ALS patients using the Single Molecule Analysis method (SIMOA) will be performed.

Research objectives comprise:

* Correlation of NfL with disease progression, including duration of ALS disease
* Correlation of NfL with the course of ALS (classic ALS or variants in the motor neuron involvement or the regional propagation patterns)
* Correlation of NfL with the progression rate of ALS

Cohorts on phenotypic variants:

The clinical phenotype of ALS will be differentiated according to the motor neuron involvement or regional propagation patterns of disease onset and clinical course.

ALS variants in relation to motor neuron involvement:

* Typical ALS: clinical features for an affection of the 1st and 2nd motor neurons are present
* Progressive muscular atrophy (PMA): only clinical features for an affection of the 2nd motor neuron are present
* Spastic ALS: predominantly clinical features for an affection of the 1st motor neuron and fewer signs of an affection of the 2nd motor neuron
* Primary lateral sclerosis (PLS): only clinical features for an affection of the 1st motor neuron are present

ALS variants in regional propagation patterns:

* Typical form: paresis of the upper or lower extremities or the bulbar region as well as the spread of the paresis to other regions
* Flail arm syndrome: primary and dominant paresis of the upper extremities and little or delayed spread of the paresis to other regions
* Flail leg syndrome: primary and dominant paresis of the lower extremities and little or delayed spread of the paresis to other regions
* Axial ALS: primary and dominant paresis of the trunk muscles and minor or delayed spread of the paresis to other regions
* Progressive bulbar paralysis: primary and dominant paresis in the bulbar region and slight or delayed spread of the paresis to other regions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of amyotrophic lateral sclerosis including specific forms
* Patient's informed consent to participate in this study
* Minimum age of 18 years
* Willingness for blood collection

Exclusion Criteria:

* Unwillingness to store and share pseudonymized medical data collected in the study
* Evaluation by the investigator, which excludes participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with clinical diagnosis of amyotrophic lateral sclerosis
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation of serum neurofilament light chain to ALS progression | 2020-2024
  correlation of serum neurofilament light chain (NfL) with the ALS progression rate as measured by the revised form of the ALS function rating scale (ALSFRS-R)
correlation of serum neurofilament light chain with ALS phenotypes | 2020-2024
  correlation of serum neurofilament light chain with ALS phenotypes in terms of type of onset and clinical variants including progressive muscle atrophy, primary lateral sclerosis, flail-arm syndrome, flail-leg syndrome and other phenotypes
correlation of serum neurofilament light chain with ALS treatment options | 2020-2024
  correlation of serum neurofilament light chain to ALS interventions such as treatment with tofersen and other medicines

SECONDARY OUTCOMES:
correlation of serum neurofilament light chain with non-pharmacologic ALS interventions | 2022-2024
  correlation of serum neurofilament light chain with non-pharmacologic ALS interventions including nutrition or ventilation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (19):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Germany (18):
  - Vivantes Klinikum Kaulsdorf, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil gGmbH, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Technische Universität Dresden, Dresden
  - Alfried Krupp von Bohlen und Halbach Krankenhaus gGmbH, Essen
  - Universitätsklinikum Essen, Essen
  - Georg-August-Universität Göttingen Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Universität Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universität Heidelberg Medizinische Fakultät Mannheim, Mannheim
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Westfälische Wilhelms-Universität Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsmedizin Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of principle investigator — https://als-charite.de/
- See also: Website of funding organization — https://canessa-als-stiftung.org/